CLINICAL TRIAL: NCT03869541
Title: Investigating the Safety of Mobilising Intensive Care Unit Patients Receiving Vasoactive Drugs: An Exploratory Observational Study
Brief Title: Exploration of Investigating ICU Mobilisation With Vasoactive Drugs
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 18SM4731
Record Dates: First submitted 2019-01-04; First posted 2019-03-11 (Actual); Results first posted 2021-09-10 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Critical Illness
Keywords: Critical Illness; Physical rehabilitation
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intensive care patients: Adult intensive care patients receiving vasoactive drugs
  Interventions: Other: Mobilization
- Intensive care unit clinicians: Clinicians for participation in a survey on the hypothetical randomization of patient participants in a future randomized controlled trial.
- ICU rehabilitation clinicians: Clinicians for participation in a survey on the feasibility of an ICU physical rehabilitation adverse event tool.

INTERVENTIONS:
Other: Mobilization — Physical rehabilitation
  Groups: Intensive care patients

SUMMARY:
There is a need to know more about the safety of mobilizing intensive care unit (ICU) patients who are receiving vasoactive drugs that support the heart and blood pressure. But before this research can be done, several uncertainties need to be addressed.

To answer these uncertainties, the investigators will ask ICU patients receiving vasoactive drugs to take part in a study in three main stages. Firstly ICU patients will be asked whether they would be happy to take part in a future research trial on the safety of mobilizing patients who are receiving vasoactive drugs. Secondly, data will be collected about the current mobilization on vasoactive drugs that occurs. Finally, the investigators will try to follow up these patients 60 days after they start the study, to carry out some questionnaires and a walking test with the patients. These tests may be used in future research to measure the effect of mobilizing patients on vasoactive drugs.

DETAILED DESCRIPTION:
The current evidence is insufficient to accurately guide clinicians to know when it is safe to start mobilizing intensive care unit (ICU) patients receiving vasoactive drugs. Before a randomized controlled trial can be designed, several uncertainties need to be addressed. This includes clarifying what standard care is, what potential recruitment rates would be and what the most suitable primary outcome measure is.

This study is an exploratory observational study which will aim to recruit up to 40 ICU patients receiving vasoactive drugs to further clarify standard care and to measure preliminary feasibility outcomes.

Upon enrolment, patients and clinicians will be surveyed about the hypothetical acceptability of recruitment into a future randomized controlled trial. Then any routine mobilization that occurs whilst the patient is receiving vasoactive drugs will be analyzed, for example, to describe how clinicians assessed safety for mobilization. Finally, patient participants will be followed up at day 60 to assess the feasibility of measuring candidate primary outcome measures.

ELIGIBILITY:
Patient participants:

Inclusion Criteria:

* Patients admitted to the ICU who are receiving vasoactive drugs.
* Age greater than or equal to 18 years old.
* Expected to remain admitted to the ICU for at least 24 hours post-enrolment.

Exclusion Criteria:

* Any patient who is expected to die imminently, as per clinical opinion.
* Any patient where mobilization is contraindicated by the nature of their existing injuries.
* Where it is clear from the medical records that participants are prisoners or offenders on probation.
* Patients with neuromuscular disease or acute brain injury or spinal cord injury.
* If the patient and/or their consultee is unable to speak English.

Clinicians participating in a survey on hypothetical randomization of patient participants:

Inclusion criteria:

* Clinicians who work in the intensive care unit where a patient participant has been admitted.

Exclusion criteria:

* None.

Clinician participants in the survey on the feasibility of the ICU physical rehabilitation adverse event tool:

Inclusion criteria:

* An ICU clinician at the research site.
* Has used the ICU physical rehabilitation adverse event tool as part of this research study.

Exclusion criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Intensive care unit patients and clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Gordon, Prof, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intensive Care Patients | Intensive Care Unit Clinicians | ICU Rehabilitation Clinicians
Started | 40 | 50 | 10
Completed | 40 | 50 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intensive Care Clinicians: Clinicians for participation in a survey on the hypothetical randomization of patient participants in a future randomized controlled trial.
- Intensive Care Rehabilitation Clinicians: Clinicians for participation in a survey on the feasibility of an ICU physical rehabilitation adverse event tool.
- Total: Total of all reporting groups
Arm/Group | Intensive Care Patients | Intensive Care Clinicians | Intensive Care Rehabilitation Clinicians | Total
Number analyzed (Participants) | 40 | 50 | 10 | 100
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Not recorded for intensive care clinicians or intensive care rehabilitation clinicians. Population: Data only collected for Intensive care patients arm for this baseline measure.
  years
    number analyzed (Participants) | 40 | 0 | 0 | 40
    (all) | 66 [54 to 72] |  |  | 66 [54 to 72]
Sex: Female, Male [Count of Participants; unit: Participants] — Not recorded for intensive care clinicians or intensive care rehabilitation clinicians. Population: Data only collected for Intensive care patients arm for this baseline measure.
  Participants
    number analyzed (Participants) | 40 | 0 | 0 | 40
    Female | 14 |  |  | 14
    Male | 26 |  |  | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not recorded for intensive care clinicians or intensive care rehabilitation clinicians. Population: Data only collected for Intensive care patients arm for this baseline measure.
  Participants
    Ethnicity: number analyzed (Participants) | 40 | 0 | 0 | 40
    Ethnicity: Black/African/Caribbean/Black British | 3 |  |  | 3
    Ethnicity: White | 29 |  |  | 29
    Ethnicity: Other / not stated | 8 |  |  | 8
Region of Enrollment [Number; unit: participants]
  United Kingdom | 40 | 50 | 10 | 100
BMI [Median (Inter-Quartile Range); unit: kg/m^2] — Not recorded for intensive care clinicians or intensive care rehabilitation clinicians. Population: Number analysed in row differs from overall due to missing data. Data only collected for Intensive care patients arm for this baseline measure.
  kg/m^2
    number analyzed (Participants) | 35 | 0 | 0 | 35
    (all) | 26 [23 to 31] |  |  | 26 [23 to 31]
APACHE (Acute physiology and chronic health evaluation)II score [Median (Inter-Quartile Range); unit: units on a scale] — A severity of disease classification system. A scale of 0 to 71, with a higher score equating to more severe disease and mortality risk.
  Not recorded for intensive care clinicians or intensive care rehabilitation clinicians. Population: Data only collected for Intensive care patients arm for this baseline measure.
  units on a scale
    number analyzed (Participants) | 40 | 0 | 0 | 40
    (all) | 16 [12 to 21] |  |  | 16 [12 to 21]
Sequential Organ Failure Assessment (SOFA) score [Median (Inter-Quartile Range); unit: units on a scale] — A score that measures the amount of organ failure. Range 0-24, increasing score = worse organ failure. Population: Data only collected for Intensive care patients arm for this baseline measure.
  units on a scale
    number analyzed (Participants) | 40 | 0 | 0 | 40
    (all) | 6 [4 to 9] |  |  | 6 [4 to 9]
Duration of invasive mechanical ventilation [Median (Inter-Quartile Range); unit: days] — Only recorded for intensive care patients arm. Population: Baseline measure only recorded for intensive care patients arm.
  days
    number analyzed (Participants) | 40 | 0 | 0 | 40
    (all) | 0 [0 to 7] |  |  | 0 [0 to 7]
Profession [Count of Participants; unit: Participants] — Profession of clinician participant. Not recorded for intensive care unit patients. Population: Data not collected for Intensive care patients arm for this baseline measure.
  Participants
    number analyzed (Participants) | 0 | 50 | 10 | 60
    Doctor |  | 17 | 0 | 17
    Nurse |  | 26 | 0 | 26
    Physiotherapist |  | 7 | 10 | 17
ICU experience [Median (Inter-Quartile Range); unit: Years] — Amount of intensive care unit experience in years. Not recorded for intensive care unit patients. Population: Missing data for two participants. Data not collected for Intensive care patients arm for this baseline measure. Data was collected for intensive care rehabilitation clinicians, however this has been summarized with a different measure type and dispersion, therefore is reported as a separate variable.
  Years
    number analyzed (Participants) | 0 | 48 | 0 | 48
    (all) |  | 11 [5 to 20] |  | 11 [5 to 20]
ICU experience of rehabilitation clinicians [Mean (Standard Deviation); unit: Years] — Population: Missing data for one participant. Data not collected for Intensive care patients arm for this baseline measure. Data was collected for intensive care clinicians arms, but summarised as a different measure type and dispersion, therefore reported as a different baseline measure.
  Years
    number analyzed (Participants) | 0 | 0 | 9 | 9
    (all) |  |  | 6 (5) | 6 (5)
Healthcare experience [Median (Inter-Quartile Range); unit: Years] — Not recorded for intensive care unit patients. Population: Missing data for two participants. Data not collected for Intensive care patients arm for this baseline measure. Data was collected for intensive care rehabilitation clinicians, however this was summarized as a different measure type and dispersion, therefore this is displayed as a separate variable.
  Years
    number analyzed (Participants) | 0 | 48 | 0 | 48
    (all) |  | 16 [9 to 26] |  | 16 [9 to 26]
Healthcare experience of rehabilitation clinicians [Mean (Standard Deviation); unit: Years] — Population: Missing data for one participant. Data not collected for Intensive care patients arm for this baseline measure. Data was collected for intensive care clinicians, however this was summarized as a different measure type and dispersion, therefore this is represented as a different baseline measure.
  Years
    number analyzed (Participants) | 0 | 0 | 9 | 9
    (all) |  |  | 9 (6) | 9 (6)

OUTCOME MEASURES:

1. Primary Outcome: Hypothetical Recruitment Rate for a Future Randomised Controlled Trial.
Description: The number of patient participants who would hypothetically accept being randomised into a future trial on the safety of mobilising patients receiving vasoactive drugs.
Time Frame: Baseline (approximately one day from enrolment)
Population: Number of participants without missing data for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 37
Participants | 30

2. Primary Outcome: Number of Participants With Follow-up at 60 Days
Description: Patient participant follow-up rate at 60 days.
Time Frame: 60 days
Population: Total number of participants in this participant group
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Participants | 40

3. Secondary Outcome: Number of Participants Rating the 'Early Versus no Rehabilitation' Randomisation Scenario Was Acceptable
Description: Survey measuring participant acceptance of hypothetical randomisation scenarios: scenario 1: early versus no rehabilitation
Time Frame: Baseline (approximately one day from enrolment)
Population: For each of the 40 patient participants, number of randomisation surveys completed by the four groups described above.
Measure: Count of Participants; unit: Participants
Groups:
- Intensive Care Patients/Consultee: Adult intensive care patients or the consultees of patients enrolled in the study.
- Intensive Care Doctors: Intensive care doctors for participation in a survey on the hypothetical randomization of patient participants in a future randomized controlled trial.
- Intensive Care Nurses: Intensive care nurses for participation in a survey on the hypothetical randomization of patient participants in a future randomized controlled trial.
- Intensive Care Physiotherapists: Intensive care physiotherapists for participation in a survey on the hypothetical randomization of patient participants in a future randomized controlled trial.
Arm/Group | Intensive Care Patients/Consultee | Intensive Care Doctors | Intensive Care Nurses | Intensive Care Physiotherapists
Number analyzed (Participants) | 37 | 32 | 34 | 40
Participants | 15 | 11 | 18 | 6

4. Secondary Outcome: Number of Participants Rating the 'Early Rehabilitation Versus Standard Care' Randomization Scenario as Acceptable
Description: Survey measuring participant acceptance of hypothetical randomization scenarios: scenario 2: early rehabilitation versus standard care
Time Frame: Baseline (approximately one day from enrolment)
Population: For each of the 40 patient participants, number of randomization surveys completed by the four groups described above.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients/Consultee | Intensive Care Doctors | Intensive Care Nurses | Intensive Care Physiotherapists
Number analyzed (Participants) | 37 | 32 | 34 | 40
Participants | 25 | 30 | 28 | 35

5. Secondary Outcome: Number of Participants Rating the 'Protocolised Rehabilitation Versus Standard Care' Randomisation Scenario as Acceptable
Description: Survey measuring participant acceptance of hypothetical randomization scenarios: scenario 3: protocolised rehabilitation versus standard care
Time Frame: Baseline (approximately one day from enrolment)
Population: For each of the 40 patient participants, number of randomisation surveys completed by the four groups described above.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients/Consultee | Intensive Care Doctors | Intensive Care Nurses | Intensive Care Physiotherapists
Number analyzed (Participants) | 36 | 32 | 35 | 40
Participants | 24 | 28 | 27 | 33

6. Secondary Outcome: Number of Participants Where Participant Pre-morbid Comorbidities Measurement Was Not Completed.
Description: Quantity of missing data resulting from measurement of participant pre-morbid co-morbidities.
Time Frame: Baseline (approximately one day from enrolment)
Population: Number of participants for whom pre-morbid evaluation of comorbidities was attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Participants | 8

7. Secondary Outcome: Number of Participants Where Participant Pre-morbid Frailty Measurements Were Not Completed.
Description: Quantity of missing data resulting from measurement of participant pre-morbid frailty.
Time Frame: Baseline (approximately one day from enrolment)
Population: Number of participants for whom pre-morbid evaluation of frailty was attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Participants | 2

8. Secondary Outcome: Number of Participants Where Participant Pre-morbid Physical Function Measurement Was Not Completed.
Description: Quantity of missing data resulting from measurement of participant pre-morbid physical function.
Time Frame: Baseline (approximately one day from enrolment)
Population: Number of participants for whom the pre-morbid measurement of physical function was attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Participants | 2

9. Secondary Outcome: Who Made the Final Decision Whether to Mobilize the Patient
Description: Recorded whenever a physiotherapist reviews a patient participant for potential physical rehabilitation whilst they are receiving vasoactive drugs and the patient was mobilized.
Time Frame: Through duration of ICU stay (average of 7 days).
Population: Number of mobilization treatments where data was available for analysis. Please note the categories presented below are not mutually exclusive e.g. a decision whether to mobilize could have been made with a nurse and a doctor. Therefore, the sum of the categories will be greater than the overall number of participants analyzed.
Measure: Number; unit: Treatment sessions
Units Other Than Participants: Treatment sessions
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Treatment sessions) | 21
Treatment sessions
  Alone | 9
  Nurse | 7
  Lead physiotherapist | 3
  Senior doctor | 1
  Doctor in charge | 4
  Surgical team | 1

10. Secondary Outcome: The Reasons for the Decision When Patient Was Mobilized.
Description: Recorded whenever a physiotherapist reviews a patient participant for potential physical rehabilitation whilst they are receiving vasoactive drugs and the patient was mobilized.
  Qualitative measure: reasons underwent content analysis, with the outcome being the themes summarizing the reasons.
Time Frame: Through duration of ICU stay (average of 7 days).
Population: Number of mobilization treatments where data was available for analysis
Measure: Number; unit: Entire group where data available
Units Other Than Participants: Entire group where data available
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Entire group where data available) | 1
Entire group where data available
  Vasoactive dose decreasing and blood pressure improved | 1
  Cardiovascularly stable and/or minimal vasoactive drug dose | 1
  Was cardiovascularly stable on initial cautious mobilisation. | 1
  Post-operative | 1
  Rationale for chest optimisation and improve strength and function. | 1
  To assess strength and alertness | 1
  Surgical wound safe to mobilise / medically stable | 1

11. Secondary Outcome: Who Made the Final Decision Whether to Not Mobilize the Patient
Description: Recorded whenever a physiotherapist reviews a patient for potential physical rehabilitation whilst they are receiving vasoactive drugs and the patient was not mobilized.
Time Frame: Through duration of intensive care stay (average 7 days)
Population: Number of reviews by a physiotherapist where patient was not mobilized and where data was available. i.e. the overall number of participants analyzed/denominator is actually the overall number of physiotherapist reviews. Please note the categories presented below are not mutually exclusive e.g. the decision not to mobilize could have been made with a nurse and a physiotherapist. Therefore, the sum of the categories exceeds with overall number of participants analyzed.
Measure: Number; unit: Reviews
Units Other Than Participants: Number of treatment reviews
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Number of treatment reviews) | 29
Reviews
  Alone | 20
  Lead physiotherapist | 6
  Nurse | 3

12. Secondary Outcome: The Reasons for the Decision When the Patient Was Not Mobilized.
Description: Recorded whenever a physiotherapist reviews a patient for potential physical rehabilitation whilst they are receiving vasoactive drugs and the patient was not mobilized.
  Qualitative variable: reasons underwent qualitative analysis, with the output of a list of themes summarizing the reasons.
Time Frame: Through duration of intensive care stay (average 7 days)
Population: Number of reviews by a physiotherapist where patient was not mobilized and where data was available.
Measure: Number; unit: Whole group where data was available
Units Other Than Participants: Whole group where data was available
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Whole group where data was available) | 1
Whole group where data was available
  Patient sedated / drowsy / confused | 1
  Patient fatigue | 1
  Patient too unwell | 1
  Blood pressure low and/or increasing/high vasoactive drug dose | 1
  Lack of staff | 1
  Pain | 1
  Did not give consent | 1
  Filter | 1

13. Secondary Outcome: The Reason Why a Mobilisation Treatment Was Stopped
Description: Recorded if a mobilisation treatment on vasoactive drugs is routinely carried out.
Time Frame: Through duration of ICU stay (average of 7 days).
Population: Number of treatment sessions for whom data was available
Measure: Number; unit: Treatments
Units Other Than Participants: Treatment sessions
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Treatment sessions) | 21
Treatments
  Aim of session achieved | 10
  Declined | 1
  Symptomatic hypotension | 2
  Patient weakness/fatigue | 6
  Pain/discomfort | 2

14. Secondary Outcome: Number of Serious Adverse Events
Description: Number of serious adverse events
Time Frame: Through whole of study, an estimated 6 months
Population: Number of mobilization treatment sessions for whom data was available
Measure: Number; unit: events
Units Other Than Participants: Treatment sessions
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Treatment sessions) | 42
events | 0

15. Secondary Outcome: Number of ICU Physical Rehabilitation Adverse Events
Description: Recorded using ICU physical rehabilitation adverse event tool, both by treating clinician and by researcher case note review.
Time Frame: Through duration of ICU stay (average of 7 days).
Population: Number of treatment sessions
Measure: Number; unit: events
Units Other Than Participants: Treatment sessions
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Treatment sessions) | 42
events
  Measured by clinicians | 3
  Measured by researchers | 6

16. Secondary Outcome: Time Taken to Complete an ICU Physical Rehabilitation Adverse Event Tool.
Description: Adverse event tool is completed if a mobilisation treatment on vasoactive drugs is routinely carried out.
Time Frame: Through duration of ICU stay (average of 7 days).
Population: Number of mobilization treatments where adverse event tool used and data available for how long it took to complete.
Measure: Number; unit: Treatments
Units Other Than Participants: Treatment sessions
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Treatment sessions) | 5
Treatments
  < 1 minute | 2
  1-3 minutes | 2
  5-10 minutes | 1

17. Secondary Outcome: Loss of Information That Occurs When Completing ICU Physical Rehabilitation Adverse Event Tool.
Description: Tool completed both by treating clinician and by researcher case note review. Number of mobilization treatment sessions on vasoactive drugs where adverse event tool is complete.
Time Frame: Through duration of ICU stay (average of 7 days).
Population: Number of mobilization treatment sessions whilst receiving vasoactive drugs
Measure: Number; unit: Treatments
Units Other Than Participants: Treatment sessions
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Number analyzed (Treatment sessions) | 42
Treatments
  Completed by clinicians | 19
  Completed by researcher | 41

18. Secondary Outcome: Feasibility and Usability of an ICU Physical Rehabilitation Adverse Event Tool Measured by Survey.
Description: A survey measuring user opinion on whether an adverse event tool was for example understandable and an appropriate length using a scale with 'yes', 'no' or 'unsure' responses. Survey adapted from Hodgson, C., Needham, D., Haines, K., Bailey, M., Ward, A., Harrold, M., Young, P., Zanni, J., Buhr, H., Higgins, A., Presneill, J. & Berney, S. 2014. Feasibility and inter-rater reliability of the ICU mobility scale. Heart Lung, 43.
Time Frame: Through second half of the study, an estimated 3 months
Population: Number of clinicians who completed the survey
Measure: Number; unit: Participants
Arm/Group | ICU Rehabilitation Clinicians
Number analyzed (Participants) | 10
Participants
  Clear, easy to understand? | 10
  Indicate its overall purpose? | 9
  Will people filling out the tool know how to? | 8
  Are the adverse events adequately defined? | 10
  Are the adverse events irrelevant or misleading? | 0
  Are the adverse events offensive or inappropriate? | 0
  Are adverse events unnecessary or repetitive? | 0
  Is the tool an appropriate length? | 10

19. Secondary Outcome: Time to First Mobilisation Treatment
Description: Number of days to first rehabilitation treatment
Time Frame: Through duration of hospital stay (average of 22 days)
Population: Number of participants with data available for this outcome.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 29
Days | 2 [1 to 7]

20. Secondary Outcome: Time to First Being Able to Sit Out of Bed.
Description: Regardless of the assistance required.
Time Frame: Through duration of hospital stay (average of 22 days)
Population: Number of patient participants with data available.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 33
Days | 5 [2 to 10]

21. Secondary Outcome: Time to First Being Able to Stand.
Description: Regardless of the assistance required.
Time Frame: Through duration of hospital stay (average of 22 days).
Population: Number of participants with data available.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 31
Days | 3 [2 to 11]

22. Secondary Outcome: Time to First Being Able to Walk.
Description: Regardless of assistance required.
Time Frame: Through duration of hospital stay (average of 22 days).
Population: Number of participants with data available.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 28
Days | 8 [4 to 21]

23. Secondary Outcome: Intensive Care Unit Length of Stay.
Time Frame: From admission to ICU discharge (an average of 7 days)
Population: Number of participants
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Days | 7 [4 to 12]

24. Secondary Outcome: Hospital Length of Stay
Time Frame: From admission to hospital discharge (average of 22 days)
Population: Number of participants
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Days | 16 [9 to 32]

25. Secondary Outcome: Intensive Care Unit Mobility Scale Level at ICU Discharge.
Description: Intensive care unit mobility scale records a patient's mobility level from 0 to 10, where 0 means no mobility and 10 means walking without assistance from people or a physical aid.
Time Frame: ICU discharge (an average of 7 days from ICU admission)
Population: Number of participants with data available.
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 38
Score on a scale | 5 [3 to 6]

26. Secondary Outcome: Number of Patient Participants Where All Candidate Primary Outcomes Are Completed.
Description: Candidate primary outcomes: mortality, health-related quality of life, disability, physical functioning questionnaire and walking test.
Time Frame: 60 days.
Population: Number of participants
Measure: Count of Participants; unit: Participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
Participants | 6

27. Secondary Outcome: The Number of Patient Participants Who Completed Each Individual Candidate Primary Outcome.
Description: as for outcome 26
Time Frame: 60 days.
Population: Number of participants
Measure: Number; unit: participants
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 40
participants
  Mortality | 40
  Health-related quality of life | 16
  Disability | 15
  Physical functioning - patient reported | 15
  Physical functioning - performance-based | 6

28. Secondary Outcome: Data to Inform a Future Sample Size for a Future Randomized Controlled Trial.
Description: Measures of central tendency and variability of data for candidate outcome measures to inform a sample size for future randomised controlled trial, e.g. physical functioning measured by the physical function domain of the RAND 36-Item Health Survey 1.0 Questionnaire (RAND SF-36 v1), scores range from 0-100, where a higher score means better physical functioning.
Time Frame: 60 days.
Population: Number of participants with data available
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Intensive Care Patients
Number analyzed (Participants) | 15
Units on a scale | 20 [0 to 50]

ADVERSE EVENTS:
Time Frame: Intensive care patients: 60 days Intensive care unit clinicians: From time of enrolment to timepoint in study where no further questionnaires were required of this study arm (length of time variable as a clinician participant could take part in one or multiple questionnaires depending if they were completing a clinical shift when a patient participant was recruited). ICU rehabilitation clinicians: From time of enrolment to time that questionnaire was returned to researcher.
Description: This study was observational (not involving changes to standard care) therefore we only monitored for and report adverse events and serious adverse events that are related to study procedures which involve contact with the participant.
Arm/Group | Intensive Care Patients | Intensive Care Unit Clinicians | ICU Rehabilitation Clinicians
All-Cause Mortality (participants affected / at risk) | 5/40 | 0/50 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/50 | 0/10
Other Adverse Events (participants affected / at risk) | 0/40 | 0/50 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03869541/Prot_SAP_000.pdf